CLINICAL TRIAL: NCT02468765
Title: Depression and Reconnaissance of Emotions in Multiple Sclerosis Patients
Brief Title: Depression and Facial Identity Recognition Abilities in Patients With Multiple Sclerosis
Acronym: SepDep
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: RC-P0040
Record Dates: First submitted 2015-06-09; First posted 2015-06-11 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis; Depression
MeSH Terms: conditions — Multiple Sclerosis; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Depressive MS patients: Neuropsychological and emotional evaluation with monitoring
  Interventions: Other: Neuropsychological and emotional evaluation with monitoring
- Non depressive MS patients: Neuropsychological and emotional evaluation with monitoring
  Interventions: Other: Neuropsychological and emotional evaluation with monitoring
- Control: Neuropsychological and emotional evaluation with monitoring
  Interventions: Other: Neuropsychological and emotional evaluation with monitoring

INTERVENTIONS:
Other: Neuropsychological and emotional evaluation with monitoring — Recognition tasks of emotional facial expressions with electroencephalogram, electrodermal activity measure and heart rate measure, questionnaires and neuropsychological tests

SUMMARY:
Cognitive and emotional disorders are often encountered in multiple sclerosis (MS) cases: depressive and bipolar disorders are twice as frequent as in general population.

Cognitive disorders, (particularly attention and dysexecutive disorders), appear in early stages of the disease's evolution, in cases of lightly or moderately disabled patients, with a recent evolution, with a "minor" form of the disease, even in Clinically Isolated Syndromes (CIS). Emotional disturbances are essentially linked to mood disorders of depression-type.

Last ten years, emotional processing in multiple sclerosis cases was investigated in various trials, especially regarding the recognition of facial and emotional expressions. These studies reported data, supporting an impairment of the perception of emotion, particularly those with negative valence.

The objective of this study is to investigate the link between recognition of facial and emotional expressions and depression in multiple sclerosis cases.

DETAILED DESCRIPTION:
Cognitive and emotional disorders in MS are common. Cognitive impairments, mainly attentional and dysexecutive, appear early in the course of the disease, in patients with mild to moderate disability, a very recent duration of evolution, a so-called "benign" form, and even in clinically isolated syndromes (CIS). Emotional disturbances mainly concern mood disorders, such as depression. Thus, Figved et al (2005) found neuropsychiatric disorders, often combined, in about 80% of their patients at the beginning of the course, with depression (59%), irritability/emotional stability (42%) and apathy (31%) being the most common. More specifically, depressive syndromes and bipolar disorders are found in MS with twice the frequency of the general population. Over the last ten years, the treatment of emotions in MS has been the subject of a few studies. MS has been the subject of several studies, notably concerning the recognition of emotional facial expressions (EFEs). Several studies have reported data in favor of an impairment of the perception of emotion perception of emotion, particularly with negative valence. These difficulties in emotion perception appear to be associated with cognitive difficulties, such as slowed processing speed and dysexecutive difficulties. This deficit appears early in the course of the disease.

Moreover, although this deficit has been little studied, such a disorder could lead to difficulties in maintaining social interaction. These patients showed a deficit in learning and recognition of non-verbal social non-verbal social cues and emotional components, independently of the cognitive impairment but more marked in the case of a functional impairment and a longer duration of the disease.

Finally, there seems to be specific relationships between problems of of emotion and poor quality of life. Indeed, the levels of certain social and psychological aspects of quality of life in MS have been correlated with these emotion perception scores, highlighting the importance of considering these emotional emotional skills in assessing the impact of MS on the patient. on the patient. The correct analysis of EFEs is a complex mental process process, requiring the functional integrity of a number of cognitive domains (working memory, attention, visual-spatial perception and executive and executive functions). In view of the impact of depression on the analytical capacities of the EFEs, described in numerous studies, the high prevalence of and alexithymia in MS patients allows us to consider these two dimensions as to consider these two dimensions as factors that may influence their identification of EFEs.

Concerning alexithymia, one study has already observed its impact on the deficit of recognition of EFEs, but no study has investigated the link between depression and such a deficiency. However, the identification of a link between the recognition abilities of EFEs and these psycho-affective disturbances would allow the development of rehabilitative treatments aiming to limit the impact of the emotional fragility of patients in their daily life and, consequently, to improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Man or Woman between 18 and 65 years old
* Participant understanding and able to speak French
* Participant understanding the Participant Informed Sheet and who has signed the Informed Consent
* Participant with Health Insurance

MS Patients :

* Patient with relapsing remitting multiple sclerosis form
* Expanded Disability Status Scale (EDSS) < 4
* Patient without motor disorders, cerebellar or significant upper limb somatosensory or visual disturbances

Control Participants :

* Participant without global cognitive deterioration

Exclusion Criteria:

* Participant taking part of other biomedical studies involving drug tests
* Participant with other neurological pathologies, head trauma with loss of consciousness, psychiatric pathologies, serious general affections, alcoholism, perception disorders, dysarthria, disorders preventing oral communication and reading, under prescription of psychotropic drugs
* Mental or visual incapacity to take part in the study
* Participant with antecedents of drug or alcohol abuse
* Allergy to the components of the gel used during the EEG
* Patients with MRI contraindications : Pacemaker or neurostimulator or Implantable Cardioverter Defibrillator (ICD), Cochlear Implants, ocular or cerebral ferromagnetic foreign body close to the nerve structures, metal prostheses,
* Uncooperative or agitated patients,
* Claustrophobic patients,
* Ventricular peritoneal shunts and neurosurgical valves,
* Braces
* MS patient without MRI in the last 4 months
* Adults under guardianship, under judicial protection, persons deprived of liberty,
* Pregnant or breast feeding women,
* MS patient with another MS form than Relapsing-Remitting,
* MS patient who encountered a relapse in the last 6 weeks,
* MS patient treated with corticoids in the last month.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Three groups will participate: Depressive MS patients, non depressive MS patients
  and a control group
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2015-04-24 (Actual); Primary Completion 2016-05-30 (Actual); Study Completion 2016-05-30 (Actual)

PRIMARY OUTCOMES:
Rate of correct answers to recognition tasks of emotional facial expressions (categorization by anger, joy or neutral) | first day of enrollement
  Rates of correct responses to the different questions of the EFEs recognition test (categorization of emotional expression (anger, joy, or neutral), assessment of the intensity of the emotion, and the degree of certainty of the responses given), compared between the three groups of participants.

SECONDARY OUTCOMES:
Correlation between facial identity recognition abilities and physiological index measured by electroencephalography | first day of enrollement
Correlation between facial identity recognition abilities and morphological index measured by magnetic resonance imaging | first day of enrollement
Correlation between facial identity recognition abilities and cognitive functions evaluated by different tests | first day of enrollement
  Correlation between facial identity recognition abilities and cognitive functions evaluated by different tests (BCcogSEP) et questionnaires (TAS 20, FIS, STAI Y et BDI II).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Hautecoeur, MD, Principal Investigator — Groupment des Hôpitaux de l'Institut Catholique de Lille
Locations (1):
- Hôpital Saint Vincent de Paul (GHICL), Lille, Hauts-de-France, France

IPD SHARING:
Plan to Share IPD: No